CLINICAL TRIAL: NCT02459847
Title: Effects of Mind-body Interventions on Stress, Anxiety, and Pain in Hand Therapy Patients
Brief Title: Mind-Body Training for Hand Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Shawn Roll, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HS-14-00320; Founders Grant (Other Grant/Funding Number: American Society of Hand Therapists)
Record Dates: First submitted 2014-11-07; First posted 2015-06-02 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Arm Injuries; Hand Injuries
MeSH Terms: conditions — Arm Injuries; Hand Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness (Experimental): Two sessions, each lasting 60-minutes total. The first session involves standard hand therapy care for the entire session. The second session begins with the participant listening to a 19-minute audio-recorded body scan (i.e., mindfulness training), followed by standard care.
  Interventions: Behavioral: Mindfulness Training; Other: Standard Care
- Biofeedback (Experimental): Two sessions, each lasting 60-minutes total. The first session involves standard hand therapy care for the entire session. The second session begins with the participant receiving 20 minutes of visual biofeedback training using sonographic imaging (i.e., sonographic biofeedback), followed by standard care.
  Interventions: Behavioral: Sonographic Biofeedback; Other: Standard Care

INTERVENTIONS:
Behavioral: Mindfulness Training
  Arms: Mindfulness
Behavioral: Sonographic Biofeedback
  Arms: Biofeedback
Other: Standard Care

SUMMARY:
The objectives of this pilot study are to: (1) evaluate acute effects of biofeedback and mindfulness training on pain, anxiety, and stress during a hand therapy visit and (2) gain understanding of patient perceptions, preferences, and experiences with mind-body interventions.

DETAILED DESCRIPTION:
Each year more than $5.7 billion is spent on outpatient therapy, which is projected to grow 6% annually over the next decade. Subsequently, healthcare reform is mandating more efficient, high-quality care to control spending. Thus, the long-term goal of this work is to develop an integrative health intervention for hand therapy that improves efficiency, enhances outcomes and reduce costs. Biofeedback and mindfulness training are two mind-body interventions that can increase patient engagement and self-efficacy. No research has investigated the integration of these mind-body interventions into treatment for hand therapy patients. This pilot research will explore the acute effects of these techniques in hand therapy patients. This study utilizes a repeated-measures crossover design with 20 participants to explore the effects of mindfulness training and the dynamic biofeedback with sonographic imaging on acute pain, anxiety, and stress. Additionally, the study will evaluate hand therapy patient preferences and perceptions of mind-body techniques. This patient-centered, clinical translational work will provide valuable feasibility data regarding the direct, acute effects of mind-body interventions to inform the development and further study of an integrative hand rehabilitation approach. This responds to a need for best practices for maximizing the mind-body connection and the call to investigate innovative uses of mindfulness to enhance patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Referral to USC Keck Hospital Hand Clinic
* Upper extremity pathology resulting in decreased hand use
* Pain with activity greater than 4 out of 10
* Scheduled to attend at least 2 therapy sessions per week
* Speak and read English
* Able to independently read and respond to questionnaires

Exclusion Criteria:

* Cast or open wounds in the distal upper extremity
* Bilateral upper extremity pathology involvement
* Significant visual or hearing deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in Salivary Cortisol throughout duration of intervention | 0, 20, 40 and 60 minutes from start of intervention session

SECONDARY OUTCOMES:
Change in State Anxiety Inventory throughout duration of intervention | 0, 20, 40 and 60 minutes from start of intervention session
Change in Visual Analogue Pain Scale throughout duration of intervention | 0, 20, 40 and 60 minutes from start of intervention session
Change from Baseline in Mindfulness Attention Awareness Scale at 2 weeks | Baseline and 2 weeks
Change from Baseline in Disabilities of the Arm, Shoulder, and Hand (DASH) Outcome Measure at 2 weeks | Baseline and 2 weeks
  The DASH Outcome Measure is a 30-item, self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb. The tool gives clinicians and researchers the advantage of having a single, reliable instrument that can be used to assess any or all joints in the upper extremity.
Change from Baseline in Five Facet Mindfulness Questionnaire - Short Form at 2 weeks | Baseline and 2 weeks
Change from Baseline in Trait Anxiety Inventory at 2 weeks | Baseline and 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shawn C Roll, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC Keck Hospital Hand Clinic, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardison ME, Roll SC. Mindfulness Interventions in Physical Rehabilitation: A Scoping Review. Am J Occup Ther. 2016 May-Jun;70(3):7003290030p1-9. doi: 10.5014/ajot.2016.018069. PMID 27089297
- [Result] Roll SC, Hardison ME, Vigen C, Black DS. Mindful Body Scans and Sonographic Biofeedback as Preparatory Activities to Address Patient Psychological States in Hand Therapy: A Pilot Study. Hand Ther. 2020 Sep;25(3):98-106. doi: 10.1177/1758998320930752. Epub 2020 Jun 9. PMID 33244321
- [Result] Takata SC, Hardison ME, Roll SC. Fostering Holistic Hand Therapy: Emergent Themes of Client Experiences of Mind-Body Interventions. OTJR (Thorofare N J). 2020 Apr;40(2):122-130. doi: 10.1177/1539449219888835. Epub 2019 Nov 25. PMID 31762376